CLINICAL TRIAL: NCT03216746
Title: Educational Methods in Oral Health for Adolescents: Influence on Knowledge and Oral Clinical Conditions
Brief Title: Oral Health Educational Methods in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Luciana Reichert Assunção Zanon, Pediatric Dentistry, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 51712315.4.0000.0102
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Adolescent Behavior
Keywords: oral health; knowledge; adolescent
MeSH Terms: conditions — Adolescent Behavior | interventions — Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral orientation and App for smartphone (Experimental): The oral health educational method of this group comprised a total of 66 adolescents aged between 14 and 19 years who received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases. The participants of this group also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Interventions: Behavioral: Oral orientation and App for smartphone
- Oral orientation (Experimental): The oral health educational method of this group comprised a total of 71 adolescents aged between 14 and 19 years who received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases.
  Interventions: Behavioral: Oral orientation
- Video orientation and App for smartphone (Experimental): The oral health educational method of this group comprised a total of 63 adolescentes aged between 14 and 19 years who received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience. The participants of this group also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Interventions: Behavioral: Video orientation and App for smartphone
- Video orientation (Experimental): The oral health educational method of this group comprised a total of 63 adolescentes aged between 14 and 19 years who received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience.
  Interventions: Behavioral: Video orientation

INTERVENTIONS:
Behavioral: Oral orientation and App for smartphone — 66 adolescents aged between 14 and 19 years. Participants enrolled in this group received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases. This intervention was carried out in a classroom, in a group with approximately 20 participants, providing an environment of discussions about the subjects covered. The duration was approximately 15 minutes. The participants also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Arms: Oral orientation and App for smartphone
Behavioral: Oral orientation — 71 adolescents aged between 14 and 19 years. Participants enrolled in this group received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases. This intervention was carried out in a classroom, in a group with approximately 20 participants, providing an environment of discussions about the subjects covered. The duration was approximately 15 minutes.
  Arms: Oral orientation
Behavioral: Video orientation and App for smartphone — 63 adolescentes aged between 14 and 19 years. Participants enrolled in this group received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience. The elaboration counted with the participation of three actors, two acting as adolescents and the third as a dental surgeon. The video had a total duration of 14 minutes. The participants also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Arms: Video orientation and App for smartphone
Behavioral: Video orientation — 63 adolescentes aged between 14 and 19 years. Participants enrolled in this group received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience. The elaboration counted with the participation of three actors, two acting as adolescents and the third as a dental surgeon. The video had a total duration of 14 minutes.
  Arms: Video orientation

SUMMARY:
Adolescence is a phase of important redefinitions and become an important period in the construction of new habits. Therefore, oral health education becomes strongly necessary, since good habits acquired at this stage may be perpetuated for adult life. The aim of this study is to evaluate the influence of an educational protocol on oral health in oral knowledge and clinical conditions in adolescence. A longitudinal study is being conducted with an initial sample of 291 adolescents enrolled in a public school in the city of Curitiba, Paraná, Brazil. The educational protocol was built in four phases. In phase I, the participants answered a questionnaire (pre-test) that included five statements about periodontal diseases and their forms of prevention. The answers were arranged in a Likert scale with a score of 1 (one) for the correct responses and 0 (zero) for the incorrect ones, obtaining, therefore, the knowledge score (KC). At this stage, adolescents is also being clinically assessed using simplified oral hygiene index (IHO-S) for dental plaque evaluation and gingival bleeding (ISG). In phase II, the sample (n = 291) is being randomly divided into two groups that receive two different educational interventions: oral orientation (OR) and video (VD). After each intervention, the questionnaire (post-test) is being reapplied. In the next phase (III), the study population (n = 291) is being again divided into four groups, and for two of them (OR + APP / VD + APP) a smartphone app was developed to messages which are being sending over a period of 30 days. In phase IV, the participants (n = 263) are answering again to the questionnaire (follow-up test) and are being reassessed clinically. Non-parametric tests and univariate and multivariate Poisson regression with robust variance will be used for statistical analysis (α = 0.05).

DETAILED DESCRIPTION:
A longitudinal study has been conducting with an initial sample of 291 adolescents enrolled in high school at a public school in the city of Curitiba, Paraná, Brazil. The educational protocol is characterized by four phases. In the first stage (Phase I), the participants are answering a questionnaire (pre-test) in order to verify the level of previous knowledge of the sample regarding periodontal diseases and their forms of prevention and are being clinically examined. In phase II the adolescents are randomly divided into two groups, which receive different educational methods: oral orientation (OR) and the application of a video (VD). After the educational interventions, the participants answer the questionnaire (post-test). In phase III, the two groups are being divided into four subgroups: oral orientation with App (OR+App), oral orientation without App (OR without App), video with App (VD+App) and video without App (VD without App). OR+App and VD+App received a mobile phone application specially developed for this study containing educational messages which are being during a period of 30 days. In the fourth phase (IV) the participants answer the questionnaire again (follow-up test) and are reassessed clinically.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of both sexes
* Regularly enrolled in the high school of a public institution

Exclusion Criteria:

* Participants with physical or mental condition
* Absence of signing consent form
* Adolescents with fixed orthodontic apparatus

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Zanon, PhD, Principal Investigator — Universidade Federal do Paraná

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vilella KD, Fraiz FC, Benelli EM, Assuncao LR. Oral Health Literacy and Retention of Health Information Among Pregnant Women: A Randomised Controlled Trial. Oral Health Prev Dent. 2017;15(1):41-48. doi: 10.3290/j.ohpd.a37712. PMID 28232973

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Orientation With App: The oral health educational method of this group comprised a total of 72 adolescents aged between 14 and 19 years who received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases. This intervention was carried out in a classroom, in a group with approximately 20 participants, providing an environment of discussions about the subjects covered. The duration was approximately 15 minutes. The participants also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Oral health educational methods: An educational protocol including different methods of education will be evaluated through the knowledge score and periodontal indexes.
- Oral Orientation Without App: The oral health educational method of this group comprised a total of 79 adolescents aged between 14 and 19 years who received standardized oral guidance performed by one of the previously trained researchers and included aspects of general and oral health and, in particular, of periodontal diseases. This intervention was carried out in a classroom, in a group with approximately 20 participants, providing an environment of discussions about the subjects covered. The duration was approximately 15 minutes. In this group, participants did not receive the App for smartphone.
  Oral health educational methods: An educational protocol including different methods of education will be evaluated through the knowledge score and periodontal indexes.
- Video With App: The oral health educational method of this group comprised a total of 68 adolescentes aged between 14 and 19 years who received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience. The elaboration counted with the participation of three actors, two acting as adolescents and the third as a dental surgeon. The video had a total duration of 14 minutes. The participants also received an App for smartphone containing messages of reinforcement in oral health which was sent during a period of 30 days.
  Oral health educational methods: An educational protocol including different methods of education will be evaluated through the knowledge score and periodontal indexes.
- Video Without App: The oral health educational method of this group comprised a total of 69 adolescentes aged between 14 and 19 years who received oral health information through an audiovisual material produced especially to this research to offer a teaching medium capable of arousing the attention of its audience. The elaboration counted with the participation of three actors, two acting as adolescents and the third as a dental surgeon. The video had a total duration of 14 minutes. In this group, participants did not receive the App for smartphone.
  Oral health educational methods: An educational protocol including different methods of education will be evaluated through the knowledge score and periodontal indexes.
Period: Overall Study
Arm/Group | Oral Orientation With App | Oral Orientation Without App | Video With App | Video Without App
Started | 72 | 79 | 68 | 69
Completed | 66 | 71 | 63 | 63
Not Completed | 6 | 8 | 5 | 6
Not completed — Lost to Follow-up | 6 | 8 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Oral Orientation Without App: This group comprised of 79 adolescents from 14 to 19 years of age who received an oral orientation from a previously trained researcher.
- Video Without App: This group comprised of 69 adolescents from 14 to 19 years of age who received a video orientation.
- Oral Orientation With App: This group comprised of 72 adolescents from 14 to 19 years of age who received an oral orientation from a previously trained researcher and also from an App developed specifically for this study.
- Video With App: This group comprised of 68 adolescents from 14 to 19 years of age who received a video orientation and also from an App developed specifically for this study.
- Total: Total of all reporting groups
Arm/Group | Oral Orientation Without App | Video Without App | Oral Orientation With App | Video With App | Total
Number analyzed (Participants) | 71 | 63 | 66 | 63 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.03 (1.158) | 16.06 (1.190) | 16.08 (1.244) | 15.98 (1.129) | 16.04 (1.175)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 33 | 40 | 145
  Male | 35 | 27 | 33 | 23 | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 71 | 63 | 66 | 63 | 263
Knowledge score [Median (Full Range); unit: score on a scale] — The knowledge score was obtained from13 statements that evaluated notions about hygiene habits and concepts of periodontal diseases. Correct answers were given a value of "1" and incorrect answers or "I don't know", score 0 (zero). Higher values represented a better outcome.
  score on a scale | 7.00 [2 to 12] | 7.00 [2 to 12] | 8.00 [3 to 11] | 7.00 [1 to 12] | 7.00 [1 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Score
Description: The knowledge score varied from 13 (five) to 0 (zero). Higher scores means better outcomes.
Time Frame: 30 days
Measure: Median (Full Range); unit: score on a scale
Groups:
- Oral Orientation: This group comprised 79 participants who received only oral orientation by a previously trained researcher.
- Oral Orientation and App: This group comprised 72 participants who received orientation through oral orientation and also an App.
- Video Orientation: This group comprised 69 adolescents who received orientation through a video.
- Video Orientation and App: This group comprised 68 adolescents who received orientation through video and also an App.
Arm/Group | Oral Orientation | Oral Orientation and App | Video Orientation | Video Orientation and App
Number analyzed (Participants) | 71 | 66 | 63 | 63
score on a scale | 11 [5 to 13] | 13 [9 to 13] | 11 [5 to 13] | 13 [10 to 13]
Statistical Analysis 1: Comparison: Oral Orientation vs Oral Orientation and App vs Video Orientation vs Video Orientation and App; Test type: Other; p = 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: The total number of "0" of participants at risk means that All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Oral Orientation Without App: This group comprised of adolescents from 14 to 19 years of age who received an oral orientation from a previously trained researcher.
- Video Without App: This group comprised of adolescents from 14 to 19 years of age who received a video orientation.
- Oral Orientation With App: This group comprised of adolescents from 14 to 19 years of age who received an oral orientation from a previously trained researcher and also from an App developed specifically for this study.
Arm/Group | Oral Orientation Without App | Video Without App | Oral Orientation With App | Video With App
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03216746/Prot_SAP_ICF_000.pdf